CLINICAL TRIAL: NCT07113197
Title: The Diagnostic Value of Duplex Ultrasound in Evaluating Infra Inguinal Arteries in Patients With Chronic Limb Threatening Ischemia : A Comparative Study With Angiography
Brief Title: Duplex Ultrasound Versus Conventional Angiography in Evaluating Lower Limb Threatening Ischemia
Acronym: DUS-CTA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Baraa Mohmamed Abdelrahman, resident doctor at sohag university hospital, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-25-7-22MS
Record Dates: First submitted 2025-08-02; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Chronic Threatening Lower Limb Ischemia
Keywords: Duplex; Angiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with chronic threatening limb ischemia (Experimental): Duplex Ultrasound (DUS) assessment of infra inguinal arterial lesions in patients with chronic threatening limb ischemia and then compared with digital subtraction angiography (DSA) as the reference standard.
  Interventions: Radiation: conventional angiography

INTERVENTIONS:
Radiation: conventional angiography — * Peak systolic velocity (PSV)
  * Velocity ratios
  * Segment visualization quality
  * Degree of stenosis

SUMMARY:
This study aims to evaluate the accuracy of Duplex Ultrasound (DUS) in assessing infra inguinal arterial lesions in patients with chronic threatening limb ischemia compared with digital subtraction angiography (DSA) as the reference standard. By comparing sensitivity, specificity, and predictive values across arterial segments, the study seeks to determine the clinical utility of DUS as a non-invasive alternative for pre-intervention vascular mapping in chronic limb-threatening ischemia.

ELIGIBILITY:
Inclusion Criteria:

- 1. Clinical diagnosis of chronic threatening lower limb ischemia (rest pain, non-healing ulcer, or gangrene).

2. Ability to provide informed consent.

Exclusion Criteria:

* 1. Hemodynamically unstable patients not fit for angiography. 2. Patients with non-atherosclerotic arterial diseases (e.g., vasculitis, Buerger's disease).

  3. Known contrast allergy or renal insufficiency precluding contrast angiography.

  4. Inadequate acoustic window or inability to undergo complete DUS examination.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-02 (Estimated); Primary Completion 2026-03-02 (Estimated); Study Completion 2026-04-02 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of DUS compared to DSA in detecting ≥50% stenosis or occlusion in femoral, popliteal, and infra popliteal arteries. | from enrollment till angioplasty (14 days mostly)
  sensitivity, specificity, positive predictive value, negative predictive value

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Sohag Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided